CLINICAL TRIAL: NCT01450631
Title: A Prospective, Randomized, Evaluation of the Prevena™ Incision Management System on Closed Incisions in Obese Subjects Undergoing Cesarean Section Surgery
Brief Title: The Use of the Prevena™ Incision Management System on Post-Surgical Cesarean Section Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AHS.2011.Prevena.Heine.03
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Post-operative Complications; Surgical Site Infection; Surgical Wound Infection
Keywords: surgical site infection; nosocomial infection; post-operative complication; surgical incision risk; surgical incision infection; negative pressure wound therapy; wound management; cesarean section surgery; wound dehiscence; wound infection; surgical closure; wound disruption; subcutaneous approximation; wound separation; seroma; hematoma; subcutaneous closure; obesity; cesarean; incision; massive obesity; obese; pregnancy; cesarean delivery; superobesity; wound complication
MeSH Terms: conditions — Surgical Wound Infection; Cross Infection; Wound Infection; Seroma; Hematoma; Obesity; Surgical Wound | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Dressing (Active Comparator): Standard-of-care includes coverage of the sutured incision with sterile gauze and non-penetrable barrier (e.g., Tegaderm™) consistent with the national standard for dressing Cesarean section incisions.
  Interventions: Device: Standard-of-care Dressing
- Prevena™ (PIMS) (Experimental): PIMS unit is a single patient use, battery-powered, disposable unit that can provide continuous -125 mmHg negative pressure over a 7-day therapy period.
  Interventions: Device: Prevena™ Incision Management System (PIMS)

INTERVENTIONS:
Device: Prevena™ Incision Management System (PIMS) — PIMS is a non-significant-risk, FDA Class II, medical device commercially available in the USA, Canada and Europe. The prospective, post-marketing clinical study described in this protocol will assess the effectiveness and functional performance of the system. The PIMS unit is a single patient use, battery-powered, disposable unit that can provide continuous -125 mmHg negative pressure over a 7-day therapy period. It is an easy to use device that also provides audible and visual alerts for low battery, maximum canister volume, and leak conditions. Additional alerts include system error and device life-cycle expiration (8 days). It is contained in a water-resistant housing, which allows the Subject to lightly shower with the device. Wound fluids are contained within the 45 mL canister.
  Other Names: PIMS; NPWT; Negative Pressure Wound Therapy
  Arms: Prevena™ (PIMS)
Device: Standard-of-care Dressing — The standard-of-care is consistent with the national standard for dressing Cesarean section incisions and includes, but not limited to, coverage of the sutured incision with sterile gauze and non-penetrable barrier (e.g., Tegaderm™). The non-penetrable barrier may be left in place for a minimum of 1 day and no longer than 2 days (± 4 hours) to promote epithelialization of the surgical incision edges. After the dressing is removed, the surgical site is left exposed to air to promote further healing. Other therapies include traditional gauze dressings with or without advanced therapies such as hydrocolloids, growth factors, and Negative Pressure Wound Therapy.
  Other Names: Standard Dressing
  Arms: Standard Dressing

SUMMARY:
The purpose of this study is to compare the post-surgical standard-of-care dressing to the Prevena™ Incision Management System in women undergoing Cesarean section surgery.

DETAILED DESCRIPTION:
This is a randomized, open-label, single-center, Phase IV, comparative interventional study looking at the effect of the Prevena™ Incision Management System (PIMS) on Cesarean section Subjects compared to a control arm treated with a standard-of-care surgical incision dressing. The prospective, post-marketing clinical study described in this protocol will assess the effectiveness and functional performance of PIMS on closed incisions. Clinical outcomes of interest for this study are defined as Surgical Site Occurrences (SSOs) that include unanticipated local inflammatory response, prolonged drainage, fluid collection, dehiscence, and surgical site infection (SSI). This investigation will compare these outcomes to a control group consisting of Subjects screened for the same inclusion and exclusion criteria but treated with a standard-of-care surgical incision dressing.

ELIGIBILITY:
Inclusion Criteria:

The Subject:

1. is a female aged ≥ 18 years
2. is able to provide her own informed consent
3. will undergo a Cesarean section procedure using a subcuticular skin closure technique within the next 42 days
4. will require a surgical incision able to be covered completely by the PIMS skin interface
5. has a BMI ≥ 35 kg/m2 as determined during the Screening Period up to 42 days pre-surgery
6. is preoperatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class I (Clean): An uninfected operative wound in which no inflammation is encountered and the respiratory, alimentary, genital, or uninfected urinary tract is not entered

      - OR -
   2. Class II (Clean Contaminated): An operative wound in which the respiratory, alimentary, genital, or uninfected urinary tract are entered under controlled conditions and without unusual contamination
7. is willing and able to return for all scheduled and required study visits
8. is not concurrently enrolled in another clinical intervention trial which may impact maternal health or the surgical site

Exclusion Criteria:

The Subject:

1. is ASA Class P4, P5, or P6 (Appendix F - American Society of Anesthesiologists (ASA) Physical Status Classification System)
2. has a systemic bacterial or fungal infection at the time of surgery
3. has a remote-site skin infection at the time of surgery
4. has a life expectancy of < 12 months
5. is preoperatively assessed to undergo a procedure with a CDC Wound Classification of:

   1. Class III (Contaminated): Open, fresh, accidental wounds, and/or major breaks in sterile technique or gross spillage from the gastrointestinal tract

      - OR -
   2. Class IV (Dirty-Infected): Old traumatic wounds with retained devitalized tissue and those that involve existing clinical infection or perforated viscera
6. experiences intraoperative hemorrhage requiring transfusion, disseminated-intravascular coagulopathy (DIC) or other medical or surgical condition during the Cesarean section deemed by the investigator to pose a prohibitively high risk for surgical re-exploration
7. who, in the investigator's opinion, would have any clinically significant condition that would impair the participant's ability to comply with the study procedures
8. has a known allergy or hypersensitivity to silver, or drape materials that contain acrylic adhesives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Heine, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for the study were recruited from a hospital Labor and Delivery Unit. Recruitment period: 26JAN2012 (site initiation) - 17DEC2013 (LPO)
Period: Overall Study
Arm/Group | Standard Dressing | Prevena™ (PIMS)
Started | 46 | 46
Completed | 43 | 42
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dressing | Prevena™ (PIMS) | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.67 (4.953) | 30.35 (5.724) | 30.01 (5.334)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 29 | 64
  White | 10 | 17 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 44 | 43 | 87
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 46.79 (5.608) | 46.25 (7.319) | 46.52 (6.489)
Gestational Age (weeks) [Mean (Standard Deviation); unit: weeks] | 37.87 (1.976) | 38.08 (1.983) | 37.97 (1.972)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Surgical Site Occurrences (SSOs) up to Day 42 (+/- 10 Days) Post Cesarean Section Surgery.
Description: Incidence of postoperative surgical site occurrences (SSOs) post Cesarean section surgery. SSOs include:
  * Unanticipated local inflammatory response
  * Prolonged drainage
  * Fluid collection
  * Dehiscence
  * Surgical site infection (SSI)
Time Frame: Post-op Day 42 (+/- 10 days) after Cesarean section surgery
Population: The Per-protocol Population was used for primary and secondary endpoint analysis.
Measure: Number; unit: participants
Arm/Group | Standard Dressing | Prevena™ (PIMS)
Number analyzed (Participants) | 43 | 39
participants | 7 | 2

2. Secondary Outcome: Incidence Rate of Surgical Incision Intervention (SII) up to Day 42 (+/- 10 Days) Post Cesarean Section Surgery.
Description: Incidence rate of surgical incision intervention (SII) post Cesarean section surgery. Interventions include:
  * Antimicrobials for surgical site infection
  * Surgical drainage of the incision
  * Surgical incision packing
  * Adjunctive negative pressure therapy
  * Debridement
  * Re-operation
Time Frame: Post-op Day: 42 (+/- 10 days) after Cesarean section surgery
Population: The Per-protocol Population was used for primary and secondary endpoint analysis.
Measure: Number; unit: participants
Arm/Group | Standard Dressing | Prevena™ (PIMS)
Number analyzed (Participants) | 43 | 39
participants | 6 | 1

ADVERSE EVENTS:
Time Frame: 1 year 10 months
Arm/Group | Standard Dressing | Prevena™ (PIMS)
Serious Adverse Events (participants affected / at risk) | 2/46 | 4/46
Other Adverse Events (participants affected / at risk) | 9/46 | 12/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dressing (N=46) | Prevena™ (PIMS) (N=46)
Cardiomyopathy (Cardiac disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Endometritis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dressing (N=46) | Prevena™ (PIMS) (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Celluitis (Infections and infestations) | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Intertrigo Candida (Infections and infestations) | 0 | 2
Mastitis (Infections and infestations) | 0 | 1
Postoperative Infection (Infections and infestations) | 3 | 1
Blister (Injury, poisoning and procedural complications) | 0 | 3
Seroma (Injury, poisoning and procedural complications) | 2 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 5 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Puritus (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days